CLINICAL TRIAL: NCT00992953
Title: The Efficacy of Virtual Reality (VR) as an Adjunct Therapy for Acute Combat-related Post-Traumatic Stress Disorder (PTSD) in Non-Combatants
Brief Title: Virtual Reality (VR) Therapy for Post-Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Office of Naval Research (ONR) (U.S. Federal Agency)
Collaborators: Naval Hospital Camp Pendleton (U.S. Federal Agency); Virtual Reality Medical Center (Unknown); United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Robert Neil McLay, Site Primary Investigator, Naval Medical Center San Diego
Organization: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-05-005
Record Dates: First submitted 2009-10-08; First posted 2009-10-09 (Estimated); Last update posted 2009-10-09 (Estimated); Status verified 2009-10

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Virtual Reality; Post Traumatic Stress Disorder; Combat; Military; Major Depressive Disorder; Anxiety; Virtual Reality Exposure with Stimulus Control; Treatment as Usual
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depressive Disorder, Major; Anxiety Disorders | interventions — Therapeutics; Virtual Reality Exposure Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality Therapy (Experimental): 10 Weeks of Virtual Reality Exposure with Stimulus Control, with up to twice a week, 90 min sessions
  Interventions: Behavioral: Virtual Reality Exposure with Stimulus Control
- Treatment As Usual (Active Comparator): Traditional Therapy and Psychiatric Medication
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Treatment as Usual — 10 weeks of therapy and/or psychiatric medication as available
  Other Names: TAU
  Arms: Treatment As Usual
Behavioral: Virtual Reality Exposure with Stimulus Control — 10 weeks of therapy, up to twice a week, 90 min sessions involving Virtual Reality Exposure with Stimulus Control
  Other Names: Virtual Reality Gradual Exposure Treatment; VRGET; Virtual Reality Exposure; VRE
  Arms: Virtual Reality Therapy

SUMMARY:
It is proposed that using Virtual Reality as part of therapy will result in improvements in Post Traumatic Stress Disorder for Service Members with PTSD related to service in Iraq and/or Afghanistan.

DETAILED DESCRIPTION:
In the treatment development phase, participants will be enrolled in Virtual Reality therapy. The therapy will be based on principals of exposure therapy, but will also incorporate aspects of physiological monitoring, and cognitive restructuring. The therapy will be modified as indicated by clinical feedback, with a fixed protocol to be developed (with length of treatment and exact methods to be used to be determined). After a fixed protocol is agreed upon, the project will enter the randomized phase. In this portion, subjects will be randomly assigned to receive either the Virtual Reality Treatment, or sent back to a waiting list during which time they will receive usual treatment. Participants will be assessed to determine which treatment (VR or treatment as usual) results in the greatest improvements in PTSD, as measured by independent assessors using the Clinician Administered PTSD scale.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Post Traumatic Stress Disorder related to military service in Iraq or Afghanistan by a Military Medical Provider.

Willing and able to give informed consent to participate Willing to give up intoxicating substances on the days of therapy

Exclusion Criteria:

* Actively suicidal, homicidal, psychotic, or having a diagnosis of alcohol dependence that does not show signs of at least early remission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2005-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Wiederhold, PhD, Principal Investigator — Virtual Reality Medical Center
Locations (2):
- United States (2):
  - Naval Hosptial Camp Pendleton, Camp Pendlton, California
  - Naval Medical Center San Diego (NMCSD), San Diego, California